CLINICAL TRIAL: NCT04481282
Title: The Combination of Terbutaline and Danazol as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-PKU010
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Terbutaline; Danazol; deanol aceglutamate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Terbutaline plus Danazol group (Experimental): Terbutaline 2.5mg tid po plus danazol 200mg bid po for 12weeks
  Interventions: Drug: Terbutaline; Drug: Danazol

INTERVENTIONS:
Drug: Terbutaline — 2.5mg po tid for 12 weeks
  Other Names: Bricanyl Brethine
Drug: Danazol — 200mg po bid for 12 weeks
  Other Names: Danocrine; Cleregil; Danol

SUMMARY:
Single-arm, open-label, single center study to assess the efficacy and safety of terbutaline plus danazol in patients with corticosteroid resistant/relapsed ITP.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a severe bleeding disorder. Approximately 2/3 of patients achieve remission from first-line therapies. However, the underlying mechanism of corticosteroid-resistant or relapsed ITP is not well understood; thus, treatment remains a great challenge. β2-AR agonist terbutaline modulates T cell differentiation and effector cell function.

A single center prospective study was performed in non-splenectomized ITP patients who were either resistant to a standard dose of corticosteroids or had relapsed. Patients were assigned to terbutaline plus danazol group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study, in order to assess the efficacy and safety of terbutaline plus danazol in patients with corticosteroid-resistant/relapsed ITP.

ELIGIBILITY:
Inclusion Criteria:

* ITP confirmed by excluding other supervened causes of thrombocytopenia;
* Platelet count of less than 30×10^9/L at enrollment;
* Patients who did not achieve a sustained response to treatment with full dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation;
* Subject has signed and dated written informed consent.
* Fertile patients must use effective contraception during treatment and observational period
* Negative pregnancy test.

Exclusion Criteria:

* Secondary immune thrombocytopenia (e.g., patients with HIV, HCV, Helicobacter pylori infection or patients with systemic lupus erythematosus)
* congestive heart failure
* severe arrhythmia
* nursing or pregnant women
* aspartate aminotransferase and alanine transaminase levels ≥ 3× the upper limit of the normal threshold criteria
* creatinine or serum bilirubin levels each 1•5 times or more than the normal range
* active or previous malignancy
* Unable to do blood routine test for the sake of time, distance, economic issues or other reasons.
* diagnosis with any of the following diseases: chronic hypertension, hyperthyroidism, diabetes, or seizure disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Sustained response | 6 months
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up. Interim analysis was scheduled at 50% through recruitment.

SECONDARY OUTCOMES:
complete remission | 6 months
  The number of participants (responders) with platelet count>=100x10^9/L (CR) and the absence of bleeding.
partial remission | 6 months
  The number of participants (responders) with platelet count >=30x10^9/L and at least a 2-fold increase in the baseline count (PR) without the administration of any other platelet increasing therapy.
time to response | 6 months
  Time to response was defined as the time from starting treatment to the time to achieve the response. Interim analysis
duration of response | 6 months
  Duration of response was measured from the achievement of response to the loss of response.
incidence of treatment-emergent adverse events | 6 months
  Adverse events were scaled according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, MD, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China